CLINICAL TRIAL: NCT01453049
Title: A Multi-center, Randomized, Double-blind, Parallel-group Study to Compare the Efficacy and Safety of Fixed-dose Rosiglitazone/Glimepiride Combination Therapy With Glimepiride Monotherapy for 24 Weeks in Drug Naive Subjects With Type 2 Diabetes
Brief Title: An Efficacy and Safety Study of Fixed-dose Rosiglitazone/Glimepiride to Treat Chinese Type 2 Diabetes Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: US FDA/EMA/SFDA decisions to rosiglitazone-containing medicines, ethic
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 113263
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2011-12

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: rosiglitazone/glimepiride, fix dose, type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- fix dose of rosiglitazone/glimepiride (Experimental): 4mg/1mg, 4mg/2mg, 4mg/4mg
  Interventions: Drug: rosiglitazone/glimepiride fix dose combination
- glimepiride (Active Comparator): 1mg, 2mg, 4mg
  Interventions: Drug: glimepiride

INTERVENTIONS:
Drug: rosiglitazone/glimepiride fix dose combination — oral, once daily, dosage is titrated according to FPG and hypoglycemia events
  Other Names: Avandaryl
  Arms: fix dose of rosiglitazone/glimepiride
Drug: glimepiride — oral, once daily, dosage is titrated according to FPG and hypoglycemia
  Other Names: Amaryl
  Arms: glimepiride

SUMMARY:
The purpose of this study is to demonstrate that the rosiglitazone/glimepiride fixed-dose combination tablet will safely and effectively control glycemia as first-line oral therapy in drug naïve subjects with type 2 diabetes. This 24-week study will compare the effects of treatment with rosiglitazone/glimepiride to treatment with glimepiride alone. The primary objective is to demonstrate superiority of rosiglitazone/glimepiride to glimepiride in lowering Glycosylated Hemoglobin (HbA1c).

DETAILED DESCRIPTION:
The antihyperglycemic effect of the thiazolidinedione (TZD) class of oral antidiabetic agents is due to their ability to increase insulin sensitivity at the cellular level, which in turn improves the ability of endogenous insulin to regulate glucose utilization by the tissues. Compounds of the sulfonylurea (SU) class act to stimulate insulin production by the pancreas, overcoming insulin resistance by increasing circulating insulin levels. The mechanisms of two kind OADs may be viewed as complementary, offering the opportunity for improved efficacy and durability of effect through coadministration of a TZD and a sulfonylurea.

Successful management of type 2 diabetes mellitus (T2DM) requires aggressive glycemic control starting at the earliest stages of the disease. Rosiglitazone/glimepiride combination therapy, with complementary mechanisms of action, has the potential to provide significant benefits over monotherapy as first line therapy. Treatment with rosiglitazone/glimepiride at this early stage of diabetes is expected to provide better glycemic control and allow a greater proportion of patients to achieve target glycemic goals than oral monotherapy.

This was a multicenter, randomized, double-blinded, parallel, study to compare the effects of treatment with rosiglitazone/glimepiride combination or glimepiride in drug naïve T2 DM patients.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* HbA1c between 7.5% and 11.0% at screening
* FPG between 7.0mmol/L and 13.3mmol/L at screening and at randomization visit
* subject was treated with diet and/or exercise alone
* QTc<450mesc or QTc<480msec for patients with bundle branch block
* Body Mass Index (BMI) >19kg/m2
* Subject has given written informed consent

Exclusion Criteria:

* Documented history of significant hypersensitivity to thiazolidinediones, sulfonylureas, or compounds with similar chemical structures
* Ongoing edema or history of edema requiring pharmacological treatment in the 12 months prior to screening
* Presence of ischemic heart disease and/or peripheral arterial disease, or NYHA grade I-IV congestive heart failure
* Taking nitrates
* Clinically significant renal or hepatic disease
* Anemia
* Severe hypertriglyceridemia (TG>=5.65mmol/L)
* Use of oral corticosteroids and Nicotinic acid
* Systolic blood pressure <170mmHg, or diastolic blood pressure > 100mmHg while on anti-hypertensive treatment
* Hyperthyroidism requiring treatment
* Diagnosed macular edema
* Women who are lactating, pregnant, or planning to become pregnant
* Presence of an active cancer or recently treated for cancer
* Drug/alcohol abuse
* Unwilling or unable to comply with the procedures described in the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- China (10):
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Suzhou, Jiangsu
  - GSK Investigational Site, Dalian, Liaoning
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Wuhan

RESULTS

PARTICIPANT FLOW:
Groups:
- Rosiglitazone+Glimepiride FDC: Fixed-dose combination (FDC) tablet of rosiglitazone (rosi) 4 milligrams (mg) and glimepiride (glim) 1 mg at Dose level 1 was administered once daily (OD) for a duration of 24 weeks (wks). In participants with fasting plasma glucose (FPG) greater than or equal to (>=) 110 mg per deciliter (dL) after 2 or 4 wks, the investigator made a blinded increase in study medication to Dose level 2 (rosi/glim, 4 mg/2 mg OD) or 3 (rosi/glim, 4 mg/4 mg OD). In any participant with hypoglycemia events at Wks 4, 8, 12, or any unscheduled visits, the dose level was reduced by one (level 3 to 2, or level 2 to 1).
- Glimepiride: Glimepiride was administered at Dose level 1 in the dose of 1 mg OD for a duration of 24 wks. In participants with FPG >=110 mg/dL after 2 or 4 wks, the investigator made a blinded increase in study medication (glim) to Dose level 2 (2 mg OD) or 3 (4 mg OD). In any participant with hypoglycemia events at Wks 4, 8, 12, or any unscheduled visits, the dose level was reduced by one (level 3 to 2, or level 2 to 1).
Period: Overall Study
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Started | 42 | 44
Completed | 1 | 2
Not Completed | 41 | 42
Not completed — Protocol Violation | 2 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawn When Sponsor Terminated Study | 35 | 36
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Randomized in Error | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride | Total
Number analyzed (Participants) | 35 | 38 | 73
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline Characteristic data are presented for all members of the Full Analysis Set, comprised of all randomized participants who received at least one dose of study medication and had at least one post-baseline efficacy assessment.
  Years | 53.6 (10.54) | 52.2 (8.57) | 52.9 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline Characteristic data are presented for all members of the Full Analysis Set, comprised of all randomized participants who received at least one dose of study medication and had at least one post-baseline efficacy assessment.
  Participants
    Female | 13 | 23 | 36
    Male | 22 | 15 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: Blood samples of participants were collected for HbA1c assessment. HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over a 2- to 3-month period. The American Diabetes Association has recommended an HbA1c value below 53 millimoles per mole (mmol/mol) (7.0%) for most participants. Change from Baseline in HbA1c was calculated as the value at Week 24 minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24
Population: Full Analysis Set (FAS): all randomized participants who received >=1 dose of study medication and had >=1 post-Baseline efficacy assessment. Missing values were imputed using Last Observation Carried Forward (used to estimate subsequent missing data points). Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent of total hemoglobin
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 38
Percent of total hemoglobin | -1.75 (1.078) | -1.47 (1.227)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 24
Description: Blood samples of participants were collected for FPG assessment. The FPG test, also known as the fasting blood sugar test, measures blood sugar levels after the participant has not eaten (fasted) for 12 to 14 hours. Change from Baseline in FBG was calculated as the value at Week 24 minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24
Population: FAS. Missing values were imputed using the Last Observation Carried Forward (LOCF) method, i.e., the last available observation was used to estimate subsequent missing data points. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 38
Millimoles per liter (mmol/L) | -1.907 (2.9601) | -0.877 (2.0673)

3. Secondary Outcome: Number of HbA1c Responders and Non-responders
Description: Blood samples of participants were collected for HbA1c assessment. HbA1c responders were defined as participants who had achieved HbA1c <7%, or who achieved a decrease of >= 0.7% from Baseline at Week 24 (LOCF).
Time Frame: Baseline (Week 0) and Week 24 (LOCF)
Population: FAS. Missing values were imputed using the LOCF method, i.e., the last available observation was used to estimate subsequent missing data points. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 38
participants
  Responders | 33 | 29
  Non-responders | 2 | 9

4. Secondary Outcome: Number of FPG Responders and Non-responders
Description: Blood samples of participants were collected for FPG assessment. FPG responders are definded as participants who had a >=1.7 mmol/L decrease from Baseline FPG or who achieved a FPG level < 6.1 mmol/L at Week 24 (LOCF).
Time Frame: Baseline (Week 0) and Week 24 (LOCF)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 38
participants
  Responders | 21 | 12
  Non-responders | 14 | 26

5. Secondary Outcome: Number of Participants Who Achieved HbA1c <7%, HbA1c <=6.5%, or Who Achieved a Decrease of >=0.7% From Baseline
Description: Blood samples of participants were collected for HbA1c assessment.
Time Frame: Baseline (Week 0) and Week 24 (LOCF)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 38
participants
  HbA1c <7% | 13 | 13
  HbA1c <=6.5% | 5 | 8
  HbA1c decrease of >=0.7% from Baseline | 33 | 29

6. Secondary Outcome: Change From Baseline in Fasting Proinsulin and Insulin at Week 24/Early Withdrawal (EW)
Description: Blood samples of participants who had fasted for 12-14 hours were collected for fasting proinsulin (precursor of insulin) and insulin assessment. Preproinsulin is sequentially processed via proinsulin, through intermediate proteolytic cleavage products, to insulin and C-peptide before release from the beta cell granule by exocytosis. Elevated levels of proinsulin are considered indicative of beta cell dysfunction. Insulin is a hormone that regulates carbohydrate and fat metabolism in the body. Change from Baseline was calculated as the value at Week 24/ EW minus the value at Baseline (Week 0).
Time Frame: Baseline (Week 0) and Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 32 | 34
Picomoles per liter (pmol/L)
  Proinsulin; n=32, 34 | -2.9 (10.18) | 3.1 (10.70)
  Insulin; n=15, 19 | 9.3 (32.27) | 24.9 (40.03)

7. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment Sensitivity (HOMA-S) at Week 24/EW
Description: Blood samples of participants who had fasted for 12-14 hours were collected for fasting glucose (FG) and insulin (FI) assessment. The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance (a condition in which natural hormone insulin becomes less effective in lowering blood sugars) and beta-cell (specialized cells in the pancreas producing insulin) function. HOMA-S is calculated using the following model to predict glucose and insulin concentrations=(FI[milliunits (mU)/milliliter (ml)]*FG [millimoles per liter (mmol/l)])/22.5. numerator, num.; denominator, denom.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio: FI*FG (num.); 22.5 (denom.)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 15 | 19
Ratio: FI*FG (num.); 22.5 (denom.) | 1.7248 (7.2543) | -2.9173 (4.5282)

8. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment Beta-cell Function (HOMA-B) at Week 24/EW
Description: Blood samples of participants who had fasted for 12 to 14 hours were collected for fasting glucose (FG) and insulin (FI) assessment. The homeostatic model assessment (HOMA) is a method used to quantify insulin resistance (a condition in which natural hormone insulin becomes less effective in lowering blood sugars) and beta-cell (specialized cells in the pancreas producing insulin) function. HOMA-B is calculated using the following mathematical model to predict glucose and insulin concentrations=(20*FI[mU/ml])/(FG[mmol/l]-3.5).
Time Frame: Baseline (Week 0) and Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio: 20*FI (num.); FG-3.5 (denom.)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 15 | 19
Ratio: 20*FI (num.); FG-3.5 (denom.) | 1.0494 (1.3229) | 1.0108 (1.1724)

9. Secondary Outcome: Number of Participants at Various Dose Levels at Week 24/EW
Description: The number of participants at the different dose levels at Week 24/EW was recorded. The different dose levels for Rosi + Glim are: Dose level 1, Rosi 4 mg + Glim 1 mg; Dose level 2, Rosi 4 mg + Glim 2 mg; Dose level 3, Rosi 4 mg + Glim 4 mg. The different dose levels for Glim are: Dose level 1, Glim 1 mg; Dose level 2, Glim 2 mg; Dose level 3, Glim 4 mg.
Time Frame: Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed. Data were missing for one participant in the rosiglitazone+glimepiride FDC arm.
Measure: Number; unit: participants
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 38
participants
  Dose Level 1 | 16 | 7
  Dose Level 2 | 8 | 18
  Dose Level 3 | 10 | 13

10. Secondary Outcome: Change From Baseline in Total Cholesterol (TC), High Density Lipoprotein-cholesterol (HDL-C), Low Density Lipoprotein-cholesterol (LDL-C), and Triglyceride (TG) at Week 24/EW
Description: Blood samples of participants who had fasted for 12 to 14 hours were collected for lipid profile (TC, HDL-C, LDL-C, TG) assessment. The lipid profile asesses the risk of heart disease. Change from Baseline in TC, HDL-C, LDL-C, and TG was calculated as the value at Week 24)/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 37
mmol/L
  TC; n=35, 36 | 0.146 (0.6736) | 0.186 (0.8849)
  HDL-C; n=35, 34 | -0.003 (0.2141) | 0.091 (0.1797)
  LDL-C; n=34, 31 | 0.002 (0.5598) | 0.067 (0.6075)
  TG; n=35, 37 | 0.344 (1.0933) | 0.056 (1.5312)

11. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen (BUN), Sodium, Potassium, Chloride, Calcium, and Phosphorus at Week 24/EW
Description: Blood samples of participants were collected for BUN and electrolyte (sodium, potassium, chloride, calcium, and phosphorus) assessment. The electrolyte balance asseses the condition of the heart and the kidneys, and BUN assesses the condition of the kidneys. Change from Baseline in BUN, sodium, potassium, chloride, calcium, and phosphorus was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population: all participants who received at least one dose of study medication. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 39 | 42
mmol/L
  BUN; n=39, 42 | 0.076 (0.8661) | 0.146 (1.3378)
  Sodium; n=39, 41 | -0.56 (2.926) | 0.33 (2.749)
  Potassium; n=39, 41 | 0.006 (0.4169) | 0.086 (0.473)
  Chloride; n=39, 41 | -1.93 (17.653) | 1.24 (3.295)
  Calcium; n=38, 35 | 0.035 (0.1481) | 0.037 (0.1122)
  Phosphorus; n=36, 35 | 0.046 (0.1315) | 0.028 (0.1980)

12. Secondary Outcome: Change From Baseline in the Ratio of TC/HDL-C and LDL-C/HDL-C at Week 24/EW
Description: Blood samples of participants who had fasted for 12 to 14 hours were collected for lipid profile (TC, HDL-C and LDL-C) assessment. The ratio of TC/HDL-C and LDL-C/HDL-C was calculated. Change from Baseline in the ratio of TC/HDL-C and LDL-C/HDL-C was calculated as the value at Week 24/EW minus the value at Baseline. For TC/HDL-C, the numerator is TC, and the denominator is HDL-C. For LDL-C/HDL-C, the numerator is LDL-C, and the denominator is HDL-C.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 33
ratio
  TC/HDL-C; n=35, 33 | 0.2295 (1.1037) | -0.1283 (0.9562)
  LDL-C/HDL-C; n=34, 31 | 0.0753 (0.8888) | -0.0782 (0.6222)

13. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (Hs-CRP) at Week 24/EW
Description: Blood samples of participants were collected for hs-CRP assessment. CRP is a marker of inflammation. High levels of CRP predict the risk of heart disease and diabetes. Change from Baseline in hs-CRP was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 37
mmol/L | -10.71 (41.368) | 2.74 (29.892)

14. Secondary Outcome: Percent Change From Baseline in High Sensitivity C-reactive Protein (Hs-CRP) at Week 24/EW
Description: Blood samples of participants were collected for hs-CRP assessment. CRP is a marker of inflammation. High levels of CRP predict the risk of heart disease and diabetes. Percent change from Baseline in hs-CRP was calculated as the value at Visit 8 (Wk 24)/ EW minus the value at Baseline divided by value at Wk 24/ EW multiplied by 100.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Full Range); unit: percent change
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 37
percent change | -39.58 [-94.8 to 2677.1] | 0.00 [-80.0 to 1320.2]

15. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D) at Week 24/EW
Description: EQ-5D is used as a measure of health outcome and includes single-item measures (coded on a 3-point scale [1, no problems; 2, some problems; 3, severe problems]) of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The instrument includes a global rating of current health using a visual analog scale (VAS): 0 (worst imaginable) to 100 (best imaginable). Health states may be converted to a single summary index by applying a formula that attaches values to each of the levels in each dimension. The index scale is -0.111 to 1. A lower index indicates worse health.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 20 | 18
scores on a scale | 0.0584 (0.1903) | 0.0447 (0.1504)

16. Secondary Outcome: Change From Baseline in Adjusted Diabetes Quality of Life (A-DQOL) Scores at Week 24/EW
Description: In diabetic participants, QOL, anxiety, and depression were measured by the A-DQOL scale . There are 46 core items (10 additional items for adolescents) and 4 major dimensions: treatment satisfaction, treatment impact, worry about long-term complications, and worry about social/vocational issues. Participants respond to all items on a 5-point Likert scale: 1, no impact, no worries, or always satisfied; 5, always affected, always worried, or never satisfied. The total score is a sum of the individual scores of all 46 items (range of 46 to 230); a lower score indicates a better QOL.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: FAS. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 17 | 16
scores on a scale | -7.0 (11.10) | -0.1 (18.63)

17. Secondary Outcome: Number of Participants With Hypoglycemic Events
Description: Blood samples of participants were collected for the assessment of blood glucose levels. Hypoglycemia is a condition that occurs when the blood glucose is below 70 mg/dL or 4 mmol/L. All participants; participants with HbA1c <7%, or who achieved a decrease of >= 0.7% from Baseline at Week 24 (HbA1c responders); and participants who had a >=1.7 mmol/L decrease from Baseline FPG or who achieved a FPG <6.1 mmol/L at Week 24 (FPG responders) were evaluated.
Time Frame: Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 40 | 43
participants
  All participants with any hypoglycemic events (HE) | 8 | 7
  HbA1c responders with any HEs | 7 | 6
  FPG responders with any HEs | 5 | 0

18. Secondary Outcome: Number of Hypoglycemic Events
Description: A hypoglycemic event is a condition that occurs when the blood glucose is below 70 mg/dL or 4 mmol/L. All participants, participants with HbA1c <7%, or who achieved a decrease of >= 0.7% from Baseline at Week 24 (HbA1c responders); and participants who had a >=1.7 mmol/L decrease from Baseline FPG or who achieved a FPG <6.1 mmol/L at Week 24 (FPG responders) were evaluated.
Time Frame: Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: Hypoglycemic events
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 40 | 43
Hypoglycemic events
  HE for all participants | 13 | 11
  HE for HbA1c responders | 12 | 10
  HE for FPG responders | 9 | 0

19. Secondary Outcome: Number of Participants With a Bone Fracture
Description: Participants with a break in the continuity (fracture) of the bone were evaluated.
Time Frame: Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 40 | 43
participants | 0 | 0

20. Secondary Outcome: Change From Baseline in White Blood Cell (WBC) Count and Platelet Count at Week 24/EW
Description: Blood samples of participants were collected for WBC count and platelet count assessment. Change from Baseline in WBC count and platelet count was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga per liter (10^9/L) cells
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 38 | 42
Giga per liter (10^9/L) cells
  WBC count | -0.418 (0.9091) | 0.148 (0.8855)
  Platelet count | -5.7 (33.73) | 3.4 (34.17)

21. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count at Week 24/EW
Description: Blood samples of participants were collected for RBC count assessment. Change from Baseline in RBC count was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Pico per liter (10^12/ L) cells
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 38 | 42
Pico per liter (10^12/ L) cells | -0.213 (0.2577) | -0.003 (0.2288)

22. Secondary Outcome: Change From Baseline in Lymphocytes, Monocytes, Neutrophils, Eosinophils, and Basophils at Week 24/EW
Description: Blood samples of participants were collected for lymphocyte, monocyte, neutrophil, eosinophil, and basophil assessment. Change from Baseline in lymphocytes, monocytes, neutrophils, eosinophils, and basophils was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: percent of WBC count
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 38 | 42
percent of WBC count
  Lymphocytes; n=38, 42 | 1.53 (5.454) | -2.33 (5.718)
  Monocytes; n=38, 42 | 0.47 (1.345) | -0.33 (1.165)
  Neutrophils; n=38, 42 | -2.84 (6.059) | 2.73 (6.065)
  Eosinophils; n=35, 42 | 0.61 (1.271) | -0.12 (1.116)
  Basophils; n=35, 42 | 0.09 (0.255) | 0.05 (0.473)

23. Secondary Outcome: Change From Baseline in Hematocrit (HCT) at Week 24/EW
Description: Blood samples of participants were collected for HCT assessment. Change from Baseline in HCT was calculated as the value at Week 24/EW minus the value at Baseline. HCT is measured as the percentage of the volume of whole blood that is made up of red blood cells.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of volume of whole blood
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 42
percentage of volume of whole blood | -1.21 (1.951) | 0.52 (2.076)

24. Secondary Outcome: Change From Baseline in Hemoglobin (HE), Mean Corpuscular Hemoglobin Concentration (MCHC), Total Protein (TP), and Albumin at Week 24/EW
Description: Blood samples of participants were collected for HE, MCHC, and TP assessment. Change from Baseline in HE, MCHC, and TP was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (G/L)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 39 | 42
Grams per liter (G/L)
  HE; n=38, 42 | -3.7 (5.81) | 1.5 (6.15)
  MCHC; n=35, 42 | -0.2 (10.05) | -0.9 (11.28)
  TP; n=39, 42 | -1.12 (3.386) | 1.45 (4.416)
  Albumin; n=39, 42 | -0.21 (2.323) | 1.44 (3.282)

25. Secondary Outcome: Change From Baseline in Mean Corpuscular Volume (MCV) at Week 24/EW
Description: Blood samples of participants were collected for MCV assessment. Change from Baseline in MCV was calculated as the value at Week 24/EW minus the value at Baseline. MCV is the average size of the red blood cells expressed in femtoliters. MCV is calculated by dividing the hematocrit (as percent) by the RBC count in millions per microliter of blood, then multiplying by 10. MCV is one of the three main RBC indices that are helpful in determining the cause of anemia.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliters (FL) per cell
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 42
Femtoliters (FL) per cell | 1.82 (2.698) | 1.01 (1.934)

26. Secondary Outcome: Change From Baseline in Mean Corpuscular Hemoglobin (MCH) at Week 24/EW
Description: Blood samples of participants were collected for MCH assessment. Change from Baseline in MCH was calculated as the value at Week 24/EW minus the value at Baseline. MCH is the average amount of hemoblobin inside a RBC expressed in picograms. MCH is calculated by dividing the hemoglobin concentration in grams per deciliter by the RBC count in millions per microliter, then multiplying by 10. MCH is one of the three main RBC indices which are helpful to determine the cause of anemia.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Picograms (pg) per cell
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 35 | 42
Picograms (pg) per cell | 0.60 (1.040) | 0.28 (0.820)

27. Secondary Outcome: Change From Baseline in Alanine Transaminase (ALT), Aspartate Aminotransferase (AST), Gamma-glutamyl Transpeptidase (GGT), Lactate Dehydrogenase (LDH), Alkaline Phosphatase (ALP), and Creatine Kinase (CK) at Week 24/EW
Description: Blood samples of participants were collected for ALT, AST, GGT, LDH, ALP, and CK assessment. Change from Baseline in ALT, AST, GGT, LDH, ALP, and CK was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 39 | 42
Units per liter (U/L)
  ALT; n=39, 42 | -6.23 (16.281) | -4.30 (12.592)
  AST; n=38, 38 | -3.5 (11.95) | -4.2 (8.67)
  GGT; n=37, 36 | -30.0 (90.40) | -1.5 (13.53)
  LDH; n=38, 37 | 2.0 (37.22) | 1.6 (23.81)
  ALP; n=38, 38 | -13.3 (13.18) | -2.8 (15.21)
  CK; n=35, 41 | 20.8 (35.85) | -1.8 (28.01)

28. Secondary Outcome: Change From Baseline in Total Bilirubin (TB), Direct Bilirubin (DB), Creatinine, and Uric Acid (UC) at Week 24/EW
Description: Blood samples of participants were collected for TB, DB, creatinine, and UC assessment. Change from Baseline in TB, DB, creatinine, and UC was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (mcmol/L)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 39 | 42
Micromoles per liter (mcmol/L)
  TB; n=39, 41 | -5.33 (5.363) | -3.44 (4.416)
  DB; n=39, 42 | -1.20 (1.923) | -0.63 (1.454)
  Creatitine; n=39, 42 | 1.03 (6.579) | -1.14 (8.239)
  UC; n=39, 42 | -13.58 (58.919) | 4.96 (60.360)

29. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Week 24/EW
Description: The blood pressure of the participants was measured. Change from Baseline in SBP and DBP was calculated as the value at Weeks 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 40 | 43
Millimeters of mercury (mmHg)
  SBP | 2.0 (15.73) | 3.1 (11.14)
  DBP | 2.2 (10.07) | 2.1 (9.73)

30. Secondary Outcome: Change From Baseline in Heart Rate at Week 24/EW
Description: The heart rate of the participants was measured. Change from Baseline in heart rate was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 40 | 43
beats per minute (bpm) | 1.1 (9.20) | -0.4 (6.96)

31. Secondary Outcome: Change From Baseline in Weight at Week 24/EW
Description: The weight of the participants was measured. Change from Baseline in weight was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 40 | 43
kilograms (kg) | 1.55 (2.632) | 1.43 (1.867)

32. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Assessment of Heart Rate at Week 24/EW
Description: Electrocardiograms of the participants were taken for the evaluation of heart rate. Change from Baseline in heart rate was calculated as the value at Week 24/EW minus the value at Baseline.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 38 | 43
bpm | -1.5 (7.65) | 3.0 (6.74)

33. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Data at Week 24/EW
Description: PR, QT, QTc, RR, QRS, and QRS axis data were measured by ECG. The PR interval (int.) starts at the beginning of the atrial contraction and ends at the beginning of the ventricular contraction. QT (QT int.) and QTc (corrected QT int.) indicate how fast the ventricles are repolarized, becoming ready for a new cycle. The RR int. represents the duration of the ventricular cardiac cycle and is an indicator of ventricular rate. QRS (QRS duration) indicates how fast the ventricles depolarize. The QRS axis is an indicator of the electrical heart axis, which is an average of all heart depolarization.
Time Frame: Baseline (Week 0) and Week 24/EW
Population: Safety Population. Only those participants contributing data at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Number analyzed (Participants) | 38 | 43
milliseconds (msec)
  PR intervals; n=38, 43 | 1.5 (9.92) | -5.6 (13.93)
  QT intervals; n=38, 43 | 3.6 (18.34) | -9.0 (31.18)
  QTc intervals; n=37, 43 | -0.9 (14.01) | -3.1 (38.14)
  RR intervals; n=37, 43 | 16.1 (80.24) | -33.4 (98.12)
  QRS intervals; n=37, 43 | -0.5 (7.52) | -1.0 (10.36)
  QRS axis intervals; n=37, 43 | 1.8 (13.17) | 0.5 (16.88)

ADVERSE EVENTS:
Description: Serious adverse events and non-serious adverse events were collected in members of the Safety Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | Rosiglitazone+Glimepiride FDC | Glimepiride
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43
Other Adverse Events (participants affected / at risk) | 6/40 | 10/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosiglitazone+Glimepiride FDC (N=40) | Glimepiride (N=43)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Dizziness (Vascular disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.